CLINICAL TRIAL: NCT05055817
Title: Development and Validation of a Clinical Risk Score to Predict the Occurrence of Bloody Stool in Hospitalized Neonates in Non-neonatal Intensive Care Unit
Brief Title: a Clinical Risk Score to Predict Bloody Stool in Neonates
Status: Withdrawn | Type: Observational
Why Stopped: no participants were included
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 2020204
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-10

CONDITIONS: Bloody Stool; Necrotizing Enterocolitis
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bloody stool group: bloody stool appear in the hospitalized neonate
  Interventions: Other: bloody stool group
- non-bloody stool group: bloody stool do not appear in the hospitalized neonate
  Interventions: Other: non-bloody stool group

INTERVENTIONS:
Other: bloody stool group — bloody stool appear in the hospitalized neonate
  Groups: bloody stool group
Other: non-bloody stool group — bloody stool do not appear in the hospitalized neonate
  Groups: non-bloody stool group

SUMMARY:
Bloody stool is a main focus in non-neonatal intensive care unit ward, and it is one of the risk factors in neonates with subsequent necrotizing enterocolitis(NEC) and usually lead to longed duration of hospitalization.

NEC is one of the most serious disease in the newborn infants, and two and more grades of NEC might lead to surgery, even death. But, it is difficult to predict when the bloody stool comes and develop to two and more grades of NEC.

DETAILED DESCRIPTION:
NEC is characterized by vomit, abdominal distention, hypoactive bowel sounds and bloody stools, even shock, disseminated intravascular coagulation(DIC) and sepsis. X-ray is shown Intestinal wall gas and/or portal vein pneumatosis and pneumoperitoneum.

Bloody stool in newborn infant is a urgent condition, and neonatologist usually need to predict whether or not two and more grades of NEC it is.

Here, the investigators will develop a score system in one retrospective cohort to predict bloody stool, and the score system is validated in another prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* more than or equal to 35 weeks' gestational age(GA)
* less than or equal to 28 days
* non-neonatal intensive care unit ward

Exclusion Criteria:

* parents' rejection
* main congenital malformation

Ages: 1 Minute to 28 Days | Sex: All
Age Groups: Child
Study Population: neonates with more than or equal to 35 weeks' GA and less than or equal to 28 days in non-neonatal intensive care unit ward are included.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
a Clinical Risk Score | up to 28 days or discharge from hospital
  a Clinical Risk Score is developed in a retrospective cohort
validation of a Clinical Risk Score | up to 28 days or discharge from hospital
  a Clinical Risk Score is validation in another prospective cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China